CLINICAL TRIAL: NCT07158658
Title: Evaluation of the Efficacy of NeoThelium FT in the Healing of Chronic Pressure Ulcers: A Prospective Case Series
Brief Title: Prospective Case Series Evaluating the Efficacy and Safety of NeoThelium FT for Chronic Pressure Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoPress
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pressure Injury
Keywords: Chronic Wounds; Wound Medicine; Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM); Cellular, Acellular, Matrix-like Product (CAMP)
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: NeoThelium FT in addition to Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoThelium FT + SOC (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT (HCT/P 361)

INTERVENTIONS:
Other: NeoThelium FT (HCT/P 361) — NeoThelium FT (HCT/P 361) is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.

SUMMARY:
This is a prospective case series evaluating the efficacy and safety of NeoThelium FT Amnion Skin Graft in the Mangement of Chronic Pressure Ulcers

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will begin SOC plus NeoThelium FT weekly applications. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of Pressure Injury/Ulcer located on the pelvis or lower extremity
3. Subject has a Pressure Injury/Ulcer Stage 2 or 3 without infection
4. Index ulcer is a minimum of 1cm2 and a maximum of 30cm2 at first treatment visit
5. Index ulcer has a depth of ≤ 1cm2, and subject is compliant to use continuous NPWT with 75-100mmHg, at the providers discretion
6. Index ulcer has a depth of > 1cm2, and subject is compliant to use continuous NPWT with 75-100mmHg
7. Pressure Injury/Ulcer is treated with offloading therapy while standing, sitting and lying down (if applicable to wound location) for 7 days prior to the first treatment visit
8. Adequate circulation of ulcer, if located on the lower extremity, demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to the first treatment visit
9. Index ulcer is free of infection prior to the first treatment visit and during screening phase.
10. Index ulcer is free of necrotic debris prior to NeoThelium FT application
11. Female subjects of childbearing potential having a negative pregnancy test prior to the first treatment visit
12. Subject is able and willing to follow the protocol requirements
13. Subject had signed informed consent
14. If 2 or more ulcers are present, the ulcers must be separated by at least 2 cm

Exclusion Criteria:

1. Subject has a known life expectancy of <1 year
2. Subject is unable to comply with protocol treatment
3. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing in the opinion of the investigator
4. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
5. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
6. Known contraindications to tissue-engineered allograft
7. Concurrent participation in alternative clinical trial that involves investigational drug or product interfering with wound treatment and/or healing
8. Subject is pregnant or breastfeeding
9. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >14 days duration within 30 days prior to the first treatment visit; or anticipated use of the above during the course of the study
10. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to the first treatment visit
11. Pressure Injury/Ulcer of Stage 4 or active osteomyelitis
12. Wound depth with visible exposed bone
13. HBOT within 14 days prior to the first treatment visit
14. Revascularization surgery on the index ulcer leg within 30 days of screening phase
15. Index ulcer suspicious of neoplasm in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-16 weeks
  Complete wound closure (100% epithelialization without drainage)

SECONDARY OUTCOMES:
Percent Area Reduction | 1-16 weeks
  Percent area reduction of wounds at 16 weeks compared to initial baseline measurement (performed using standardized methods of wound area measurement)
Wound Closure | 2 weeks
  Evaluate wounds remaining closed for the 2 week follow
Number of Grafts | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Chair — SygNola, LLC
Locations (1):
- MedCentris of Bossier City, Bossier City, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No